CLINICAL TRIAL: NCT05236686
Title: A Prospective, Multi-center, Single-Arm Phase II Clinical Study to Evaluate Safety and Effectiveness of Hepato-celiac Lymphadenectomy in the Treatment of Advanced and Recurrent Ovarian Cancer
Brief Title: Survival Effect of Hepato-celiac Lymphadenectomy In Primary or Relapsed Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zsfud-GynOncol-005
Record Dates: First submitted 2022-01-28; First posted 2022-02-11 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Ovarian Cancer; Surgery; Lymph Node Metastasis; Hepato-celiac Lymphadenectomy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepato-celiac lymphadenectomy (Experimental): This single-arm, multi-center, phase II trial is to evaluate the safety and effectiveness of hepato-celiac lymphadenectomy in the treatment of ovarian cancer with hepato-celiac lymph nodes metastases, in the circumstance of primarily diagnosed advanced epithelial ovarian cancer (primary debulking surgery or interval debulking surgery) and of platinum-sensitive recurrent ovarian cancer (no more than 4 lines of therapy).
  Interventions: Procedure: Hepato-celiac lymphadenectomy

INTERVENTIONS:
Procedure: Hepato-celiac lymphadenectomy — Hepato-celiac lymphadenectomy in the treatment of epithelial ovarian cancer, with a maximum cytoreduction, in the circumstance of primarily diagnosed advanced epithelial ovarian cancer (primary debulking surgery or interval debulking surgery) and of platinum-sensitive recurrent ovarian cancer (no more than 4 lines of therapy).

SUMMARY:
The purpose of this study is to evaluate the safety and the effectiveness of hepato-celiac lymphadenectomy in the treatment of primarily diagnosed advanced epithelial ovarian cancer and platinum-sensitive recurrent ovarian cancer.

DETAILED DESCRIPTION:
This single-arm, multi-center, phase II trial is to evaluate the safety and effectiveness of hepato-celiac lymphadenectomy in the treatment of ovarian cancer with hepato-celiac lymph nodes metastases, in the circumstance of primarily diagnosed advanced epithelial ovarian cancer (primary debulking surgery or interval debulking surgery) and of platinum-sensitive recurrent ovarian cancer (no more than 4 lines of therapy).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years to ≤ 75 years.
* Pathologic confirmed stage III or IV epithelial ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma (EOC, PPC, FTC) or platinum sensitive, relapsed EOC, PPC or FTC (no more than 4 lines of therapy)
* Hepato-celiac lymph nodes metastases diagnosed by imaging before surgery and enlarged palpable lymph nodes by surgical findings
* Assessed by the experienced surgeons, complete resection is feasible according to preoperative evaluation
* 1 to 3 episodes of neoadjuvant chemotherapy is allowed in primary settings
* Platinum sensitive relapse is defined as those with platinum-free interval of 6 months or more.
* ASA score of 1 to 2
* ECOG performance status of 0 to 2
* Adequate bone marrow, liver and renal function to receive chemotherapy and subsequently to undergo surgery:
* White blood cells >3,000/µL, absolute neutrophil count ≥1,500/µL, platelets ≥100,000/µL, hemoglobin ≥9 g/dL,
* Serum creatinine <1.25 x upper normal limit (UNL) or creatinine clearance ≥60 mL/min according to Cockcroft-Gault formula or to local lab measurement
* Serum bilirubin <1.25 x UNL, AST(SGOT) and ALT(SGPT) <2.5 x UNL
* Comply with the study protocol and follow-up.
* Written informed consent.

Exclusion Criteria:

* Patients with non-epithelial ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma.
* Low-grade carcinoma.
* Mucinous ovarian cancer.
* Infeasible complete resection according to preoperative evaluation
* Unresectable pulmonary and hepatic parenchymal metastases, multiple thoracic lymph nodes metastases, brain or bone metastases according to preoperative evaluation.
* Carcinomatosis on small bowel mesentery or intestinal wall by surgical findings and infeasible optimal surgery by bowel resection or peritonectomy.
* Progression after neoadjuvant chemotherapy in primary settings.
* Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ or breast cancer (without any signs of relapse or activity).
* Any other concurrent medical conditions contraindicating surgery or chemotherapy that could compromise the adherence to the protocol.
* Other conditions, such as religious, psychological and other factors, that could interfere with provision of informed consent, compliance to study procedures, or follow-up.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
2-years Non-Progression Rate | Participants will be followed up to 2 years after randomization
  The proportion of patients without disease progression or death at 2 years after entry into the study.

SECONDARY OUTCOMES:
Progression free survival | Participants will be followed up to 24 months after randomization
  The time from entry into the study to the diagnosis of the first progression or recurrence or death, whichever occurs first
Overall survival | Participants will be followed up to 60 months after randomization
  The time from date of randomization until the date of death from any cause or last follow-up
Objective response rate | Participants will be followed up to 24 months after randomization
  The proportion of patients who achieved complete response (CR) or partial response (PR)
Disease control rate | Participants will be followed up to 24 months after randomization
  The proportion of patients who achieved complete response (CR) or partial response (PR) or stable disease (SD)
Post-operative complications | Participants will be followed up to 90 days after randomization
  Postoperative 30-day, 60-day and 90-day complications
Quality of life assessments (QLQ-C30) | Baseline; 6 months, 12 months and 24 months after randomization
  Assessment of potential impact of first line treatment on functionality and well-being in patients by the EORTC core quality of life questionnaire (QLQ-C30, version 3.0).
Quality of life assessments (FACT-Q) | Baseline; 6 months, 12 months and 24 months after randomization
  Assessment of potential impact of first line treatment on functionality and well-being in patients by functional assessment of cancer therapy-ovary (FACT-O, version 4).
Patterns of subsequent recurrence | Participants will be followed up to 24 months after randomization
  The number and sites of subsequent recurrence, including pelvic, abdominal, retroperitoneal lymph nodes, hepato-celiac lymph nodes and distant metastases and ascites, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Rongyu Zang, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No